CLINICAL TRIAL: NCT01147744
Title: A Randomised Double-Blind, Double-Dummy, Placebo-Controlled, Stratified, Parallel-Group, Multicentre, Dose Ranging Study to Evaluate the Efficacy and Safety of GSK2190915 Tablets Administered Once Daily, Fluticasone Propionate Inhalation Powder 100mcg Twice Daily and Montelukast 10mg Once Daily Compared With Placebo for 8 Weeks in Adolescent and Adult Subjects With Persistent Asthma While Treated With Short Acting Beta2-agonist.
Brief Title: Dose Ranging Study Evaluating the Efficacy and Safety of GSK2190915 Administered Once Daily
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112186
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: Efficacy; Asthma; Safety; Fluticasone Propionate; FLAP; Beta-agonists; GSK2190915; Montelukast; Placebo; FLAIR
MeSH Terms: conditions — Asthma | interventions — Fluticasone; 3-(3-tert-butylsulfanyl-1-(4-(6-ethoxypyridin-3-yl)benzyl)-5-(5-methylpyridin-2-ylmethoxy)-1H-indol-2-yl)-2,2-dimethylpropionic acid; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- GSK2190915 10mg and placebo (Experimental): GSK2190915 10mg (1 x 10mg, 1 x placebo tablets) once daily in the morning and placebo caspule once daily in the evening and inhaled placebo twice daily via ACCUHALER/DISKUS
  Interventions: Drug: GSK2190915 10mg; Drug: Placebo GSK2190915 one tablet; Drug: Placebo montelukast; Drug: Placebo fluticasone propionate via ACCUHALER/DISKUS
- GSK2190915 30mg and placebo (Experimental): GSK2190915 30mg (1 x 30mg, 1 x placebo tablets) once daily in the morning and placebo caspule once daily in the evening and inhaled placebo twice daily via ACCUHALER/DISKUS
  Interventions: Drug: GSK2190915 30mg; Drug: Placebo GSK2190915 one tablet; Drug: Placebo montelukast; Drug: Placebo fluticasone propionate via ACCUHALER/DISKUS
- GSK2190915 100mg QD and placebo (Experimental): GSK2190915 100mg (1 x 100mg, 1 x placebo tablets) once daily in the morning and placebo caspule once daily in the evening and inhaled placebo twice daily via ACCUHALER/DISKUS
  Interventions: Drug: GSK2190915 100mg; Drug: Placebo GSK2190915 one tablet; Drug: Placebo montelukast; Drug: Placebo fluticasone propionate via ACCUHALER/DISKUS
- GSK2190915 300mg QD and placebo (Experimental): GSK2190915 300mg (1 x 100mg, 1 x 200mg tablets) once daily in the morning and placebo caspule once daily in the evening and inhaled placebo twice daily via ACCUHALER/DISKUS
  Interventions: Drug: GSK2190915 300mg; Drug: Placebo montelukast; Drug: Placebo fluticasone propionate via ACCUHALER/DISKUS
- Fluticasone propionate 100mcg and placebo (Active Comparator): Fluticasone propionate 100mcg twice daily via ACCUHALER/DISKUS and two placebo tablets in the morning and one placebo capsule in the evening
  Interventions: Drug: Fluticasone Propionate 100mcg via ACCUHALER/DISKUS; Drug: Placebo montelukast; Drug: Placebo GSK2190915 two tablets
- Montelukast 10mg and placebo (Active Comparator): Montelukast 10mg (1 x 10mg capsule) once daily in the evening and two placebo tablets in the morning and inhaled placebo twice daily via ACCUHALER/DISKUS
  Interventions: Drug: Montelukast 10mg; Drug: Placebo fluticasone propionate via ACCUHALER/DISKUS; Drug: Placebo GSK2190915 two tablets
- Placebo Comparator (Placebo Comparator): Two GSK2190915 placebo tablets once daily in the morning, montelukast placebo capsule once daily in the evening and fluticasone propionate placebo twice daily via ACCUHALER/DISKUS
  Interventions: Drug: Placebo montelukast; Drug: Placebo fluticasone propionate via ACCUHALER/DISKUS; Drug: Placebo GSK2190915 two tablets

INTERVENTIONS:
Drug: Fluticasone Propionate 100mcg via ACCUHALER/DISKUS — Fluticasone propionate 100mcg twice daily via ACCUHALER/DISKUS
  Arms: Fluticasone propionate 100mcg and placebo
Drug: GSK2190915 100mg — GSK2190915 100mg (1 x 100mg) once daily in the morning
  Arms: GSK2190915 100mg QD and placebo
Drug: GSK2190915 10mg — GSK2190915 10mg (1 x 10mg) once daily in the morning
  Arms: GSK2190915 10mg and placebo
Drug: GSK2190915 300mg — GSK2190915 300mg (1 x 100mg, 1 x 200mg tablets) once daily in the morning
  Arms: GSK2190915 300mg QD and placebo
Drug: GSK2190915 30mg — GSK2190915 30mg (1 x 30mg) once daily in the morning
  Arms: GSK2190915 30mg and placebo
Drug: Montelukast 10mg — Montelukast 10mg (1 x 10mg capsule) once daily in the evening
  Arms: Montelukast 10mg and placebo
Drug: Placebo GSK2190915 one tablet — Placebo tablet, one tablet once daily in the morning
  Arms: GSK2190915 100mg QD and placebo; GSK2190915 10mg and placebo; GSK2190915 30mg and placebo
Drug: Placebo montelukast — Placebo capsule once daily in the evening
  Arms: Fluticasone propionate 100mcg and placebo; GSK2190915 100mg QD and placebo; GSK2190915 10mg and placebo; GSK2190915 300mg QD and placebo; GSK2190915 30mg and placebo; Placebo Comparator
Drug: Placebo fluticasone propionate via ACCUHALER/DISKUS — Inhaled placebo twice daily via ACCUHALER/DISKUS
  Arms: GSK2190915 100mg QD and placebo; GSK2190915 10mg and placebo; GSK2190915 300mg QD and placebo; GSK2190915 30mg and placebo; Montelukast 10mg and placebo; Placebo Comparator
Drug: Placebo GSK2190915 two tablets — Placebo tablet, two tablets once daily in the morning
  Arms: Fluticasone propionate 100mcg and placebo; Montelukast 10mg and placebo; Placebo Comparator

SUMMARY:
To evaluate the efficacy, dose response and safety of four doses of GSK2190915 in tablet form (10mg, 30mg, 100mg and 300mg) administered once daily, over 8 weeks compared with placebo in adolescent and adult subjects (12 years of age and older) with persistent asthma. These data will form the basis for the selection of the optimal daily dose of GSK2190915 to be carried forward in Phase III asthma studies. The study also includes Fluticasone Propionate Inhalation Powder (100 mcg, twice daily) and Montelukast (10mg, once daily) to allow for an exploratory analysis of the efficacy of GSK2190915 versus a low dose inhaled corticosteroid and a leukotriene receptor antagonist.

ELIGIBILITY:
Inclusion Criteria:

* Type of Subject: Outpatient
* Age: ≥12 years of age
* Gender: Eligible Female (females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control)
* Asthma Diagnosis: As defined by NIH
* Severity of Disease: FEV1 50-85% predicted AND in current and former smokers a post salbutamol/albuterol ratio >0.70
* Reversibility: ≥12% and ≥200mL in FEV1 within 30 ±15 minutes following salbutamol/albuterol
* Current anti-asthma therapy: Using short-acting beta-agonist (SABA) for ≥3 months
* Tobacco use: Non-smoker /former smoker with ≤10 pack years or current smoker with ≤10 pack years
* QTC: QTc(F)<450msec or QTc(F)<480 for subjects with Bundle Branch Block
* Liver function: Normal liver function
* Informed Consent

Exclusion Criteria:

* History of Life-threatening asthma: Within previous 5 years
* Asthma Exacerbation: Requiring OCS within 3 months or hospitalisation within 6 months
* Respiratory Infection: Not resolved within the 4 weeks before V1 AND led to a change in asthma management OR treatment with antibiotics OR is expected to affect the subject's asthma status or ability to participate
* Corticosteroid Use: ICS used within 6 weeks or OCS/depot corticosteroids within 12 weeks
* OATP1B1 substrates: OATP1B1 substrates (e.g. statins, rifampicin, bromosulphophthalein, benzylpenicillin, methotrexate) within 4 weeks
* Immunosuppressive medications: Either using or required during the study
* Liver disease: Current or chronic history
* Concurrent disease/abnormalities: Clinically significant uncontrolled disease
* Investigational medications: Participation in a study or used investigational drug within 30 days
* Drug allergy: β-agonists, corticosteroids, constituents of inhalers
* Milk Protein Allergy: History of severe milk protein allergy
* Compliance: Factors likely to impair compliance either with regards to study medication, procedures or attendance
* Unable or unwilling to follow instructions: Procedures, dosing directions, e-diaries or pMDIs
* History of alcohol or drug abuse: Likely to interfere with the study
* Affiliation with Investigator's Site: Relative or employee

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2010-06-28 (Actual); Primary Completion 2011-10-06 (Actual); Study Completion 2011-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (58):
- United States (22):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Bellingham, Washington
- Bulgaria (6):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Varna
- Japan (8):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- Poland (7):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Libiąż
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Tarnów
- Romania (5):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Timișoara
- Ukraine (10):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Yalta
  - GSK Investigational Site, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Follows RM, Snowise NG, Ho SY, Ambery CL, Smart K, McQuade BA. Efficacy, safety and tolerability of GSK2190915, a 5-lipoxygenase activating protein inhibitor, in adults and adolescents with persistent asthma: a randomised dose-ranging study. Respir Res. 2013 May 17;14(1):54. doi: 10.1186/1465-9921-14-54. PMID 23682661
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 112186 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112186 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112186 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112186 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112186 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112186 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112186 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1245 participants were screened, of these, 363 participants failed screening, 882 entered the run-in phase and a total of 700 participants were randomized and included in Intent to Treat (ITT) Population . The study was conducted from 28 Jun 2010 to 06 October 2011, in the Ukraine, United States, Bulgaria, Poland, Japan, Romania.
Pre-assignment Details: Participants were screened (Visit 1) for eligibility, which included reversibility testing. Following screening and a 14-days Run-in Period, participants who met the eligibility criteria for randomization to study treatment at Visit 3 were randomly assigned to receive one of seven double-blind treatments for 8 weeks.
Groups:
- Placebo: Participants received two tablets of placebo orally plus one dose of fluticasone propionate (FP) matching placebo twice daily (BID) via dry powder inhaler (DPI) in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast matching placebo orally once daily (QD) in evening for the 8-Weeks.
- GSK2190915 10 Milligrams (mg): Participants received one tablet of 10 mg GSK2190915 orally QD and one tablet of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- GSK2190915 30mg: Participants received one tablet of 30 mg GSK2190915 orally QD and one tablet of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- GSK2190915 100mg: Participants received one tablet of 100 mg GSK2190915 orally QD and one tablet of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- GSK2190915 300mg: Participants received one tablet of 100 mg GSK2190915 and one tablet of 200 mg GSK 2190915 orally QD plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo BID via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- Fluticasone Propionate 100 Microgram (mcg): Participants received one dose of FP 100 mcg BID via DPI plus two tablets of placebo in morning and another dose of FP 100 mcg via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- Montelukast 10mg: Participants received two tablets of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast 10 mg orally QD in evening for the 8-Weeks.
Period: Overall Study
Arm/Group | Placebo | GSK2190915 10 Milligrams (mg) | GSK2190915 30mg | GSK2190915 100mg | GSK2190915 300mg | Fluticasone Propionate 100 Microgram (mcg) | Montelukast 10mg
Started | 100 | 99 | 100 | 100 | 101 | 103 | 97
Completed | 71 | 76 | 82 | 82 | 76 | 83 | 78
Not Completed | 29 | 23 | 18 | 18 | 25 | 20 | 19
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 1 | 3 | 1
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 11 | 11 | 9 | 11 | 13 | 8 | 7
Not completed — Adverse Event | 1 | 2 | 3 | 0 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 8 | 4 | 2 | 2 | 2 | 5 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor decision to amend protocol | 7 | 4 | 2 | 5 | 7 | 2 | 6
Not completed — Met Protocol-defined Stopping Criteria | 1 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received two tablets of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- GSK2190915 10 mg: Participants received one tablet of 10 mg GSK2190915 orally QD and one tablet of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- GSK2190915 30 mg: Participants received one tablet of 30 mg GSK2190915 orally QD and one tablet of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- GSK2190915 100 mg: Participants received one tablet of 100 mg GSK2190915 orally QD and one tablet of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- GSK2190915 300 mg: Participants received one tablet of 100 mg GSK2190915 and one tablet of 200 mg GSK 2190915 orally QD plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo BID via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- Fluticasone Propionate 100 mcg: Participants received one dose of FP 100 mcg BID via DPI plus two tablets of placebo in morning and another dose of FP 100 mcg via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
- Montelukast 10 mg: Participants received two tablets of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast 10 mg orally QD in evening for the 8-Weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 30 mg | GSK2190915 100 mg | GSK2190915 300 mg | Fluticasone Propionate 100 mcg | Montelukast 10 mg | Total
Number analyzed (Participants) | 100 | 99 | 100 | 100 | 101 | 103 | 97 | 700
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (16.13) | 40 (15.56) | 43.1 (16.17) | 42.2 (14.63) | 42.2 (14.15) | 41.5 (15.16) | 44.3 (14.97) | 42.2 (15.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 91 | 94 | 92 | 93 | 97 | 89 | 644
  Male | 12 | 8 | 6 | 8 | 8 | 6 | 8 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 4
  Asian | 12 | 13 | 12 | 11 | 13 | 12 | 12 | 85
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 12 | 10 | 9 | 9 | 7 | 9 | 62
  White | 82 | 74 | 78 | 78 | 78 | 83 | 76 | 549
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to the End of the 8-Week Treatment Period in Trough Forced Expiratory Volume in One Second (FEV1)
Description: Pulmonary function was measured by forced expiratory volume in one second, defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is defined as the morning (AM) pre-dose and pre-rescue bronchodilator FEV1 at the clinic visit. Baseline was the pre-dose value obtained at Visit 3. Change from Baseline was calculated as the end of Week 8 value minus the Baseline value. Analysis of covariance (ANCOVA) model used for statistical analysis. ITT Population was comprised of all participant randomized to treatment who received at least one dose of double-blind study medication.
Time Frame: Baseline and Week 8
Population: ITT population. When possible, data from participants who withdrew prematurely from the study were included in the analyses. Any evaluable subject whose FEV1 measurement at Week 8 was missing was included in the analysis by imputation, using the preceding non-missing FEV1 value (last observation carried forward [LOCF]).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 30 mg | GSK2190915 100 mg | GSK2190915 300 mg | Fluticasone Propionate 100 mcg | Montelukast 10 mg
Number analyzed (Participants) | 98 | 96 | 99 | 100 | 98 | 100 | 95
Liters | 0.12 (0.04) | 0.18 (0.04) | 0.23 (0.04) | 0.19 (0.04) | 0.19 (0.04) | 0.31 (0.04) | 0.19 (0.04)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; Test type: Superiority or Other; p = 0.326, ANCOVA — The study type I error rate was controlled at 5% level for primary efficacy analyses using the Week 8 trough FEV1 endpoint, by performing statistical tests of GSK2190915 versus placebo, sequentially from highest dose (300 mg) to lowest dose (10 mg); ANCOVA model used with covariates of Baseline trough FEV1, age, gender, country and smoking status. The LOCF method used to impute missing data; Mean Difference (Net) = 0.056, 95% CI 2-sided [-0.06 to 0.17]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30 mg; Test type: Superiority or Other; p = 0.066, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.104, 95% CI 2-sided [-0.01 to 0.22]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100 mg; Test type: Superiority or Other; p = 0.224, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.069, 95% CI 2-sided [-0.04 to 0.18]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300 mg; Test type: Superiority or Other; p = 0.271, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.062, 95% CI 2-sided [-0.05 to 0.17]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.189, 95% CI 2-sided [0.08 to 0.30]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10 mg; Test type: Superiority or Other; p = 0.220, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.070, 95% CI 2-sided [-0.04 to 0.18]

2. Secondary Outcome: Mean Change From Baseline in Daily Evening (PM) Peak Expiratory Flow (PEF) Averaged Over the 8-Week Treatment Period
Description: Peak expiratory flow is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Change from Baseline was calculated as the value of the averaged PEF daily (pre-dose and pre-rescue bronchodilator) evening over the 8-Week treatment period minus the Baseline value (defined as the last 7 days prior to randomization of the participants)
Time Frame: Baseline up to Week 8
Population: ITT Population. Only those participants with analyzable data at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 30 mg | GSK2190915 100 mg | GSK2190915 300 mg | Fluticasone Propionate 100 mcg | Montelukast 10 mg
Number analyzed (Participants) | 99 | 99 | 99 | 100 | 101 | 101 | 97
Liters per minute | 8.01 (3.19) | 7.62 (3.19) | 9.37 (3.20) | 6.21 (3.17) | 10.33 (3.15) | 10.46 (3.16) | 8.53 (3.24)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; Test type: Superiority or Other; p = 0.932, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = -0.385, 95% CI 2-sided [-9.25 to 8.48]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30 mg; Test type: Superiority or Other; p = 0.762, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = 1.367, 95% CI 2-sided [-7.50 to 10.23]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100 mg; Test type: Superiority or Other; p = 0.689, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Median Difference (Net) = -1.798, 95% CI 2-sided [-10.62 to 7.03]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300 mg; Test type: Superiority or Other; p = 0.605, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = 2.321, 95% CI 2-sided [-6.49 to 11.13]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.584, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = 2.460, 95% CI 2-sided [-6.36 to 11.28]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10 mg; Test type: Superiority or Other; p = 0.907, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = 0.529, 95% CI 2-sided [-8.40 to 9.45]

3. Secondary Outcome: Mean Change From Baseline in Daily Trough AM PEF Averaged Over the 8-Week Treatment Period
Description: The PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Trough AM PEF is defined as the AM pre-dose and pre-rescue bronchodilator at the clinic visit. Change from Baseline was calculated as the value of the averaged PEF daily (pre-dose and pre-rescue bronchodilator) AM over the 8-Week treatment period minus the Baseline value (defined as the last 7 days prior to randomization of the participants).
Time Frame: Baseline up to Week 8
Population: ITT Population. Only those participants with analyzable data at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 30 mg | GSK2190915 100 mg | GSK2190915 300 mg | Fluticasone Propionate 100 mcg | Montelukast 10 mg
Number analyzed (Participants) | 99 | 99 | 99 | 100 | 101 | 100 | 97
Liters per minute | 11.77 (3.28) | 13.23 (3.28) | 15.52 (3.29) | 8.72 (3.26) | 16.35 (3.24) | 15.25 (3.26) | 17.38 (3.32)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; Test type: Superiority or Other; p = 0.753, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = 1.463, 95% CI 2-sided [-7.65 to 10.58]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30 mg; Test type: Superiority or Other; p = 0.419, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = 3.750, 95% CI 2-sided [-5.36 to 12.87]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100 mg; Test type: Superiority or Other; p = 0.510, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = -3.046, 95% CI 2-sided [-12.12 to 6.03]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300 mg; Test type: Superiority or Other; p = 0.320, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = 4.585, 95% CI 2-sided [-4.47 to 13.64]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.452, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = 3.484, 95% CI 2-sided [-5.61 to 12.58]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10 mg; Test type: Superiority or Other; p = 0.229, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline trough PM PEF, age, gender, country and smoking status; Mean Difference (Net) = 5.615, 95% CI 2-sided [-3.55 to 14.78]

4. Secondary Outcome: Mean Change From Baseline in the Percentage of Symptom-free Days Averaged Over the 8-Week Treatment Period
Description: Asthma symptoms were recorded in a daily electronic diary (eDiary) by the participants every day in the evening at bedtime and before taking any rescue or study medication and before the assessment of the PEF measurement. Participant's responses to evening assessments indicated no symptoms were considered to be symptom free. For participants, the symptom free days were assessed during the 8-Week treatment period. Change from Baseline was calculated as the averaged of symptom-free days during the 8-Week treatment period minus the Baseline value. Baseline was defined as the last 7 days prior to randomization of the participants.
Time Frame: Baseline up to Week 8
Population: ITT Population. Endpoint obtained from the daily diary record used all available data over the period of interest. No imputations were performed on missing data from the daily diary record.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free days
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 30 mg | GSK2190915 100 mg | GSK2190915 300 mg | Fluticasone Propionate 100 mcg | Montelukast 10 mg
Number analyzed (Participants) | 99 | 99 | 99 | 100 | 101 | 101 | 97
Percentage of symptom-free days | 13.98 (2.84) | 15.15 (2.84) | 18.54 (2.84) | 15.31 (2.82) | 14.06 (2.81) | 22.18 (2.81) | 16.87 (2.87)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; Test type: Superiority or Other; p = 0.771, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 1.169, 95% CI 2-sided [-6.73 to 9.07]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30 mg; Test type: Superiority or Other; p = 0.257, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 4.560, 95% CI 2-sided [-3.33 to 12.45]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100 mg; Test type: Superiority or Other; p = 0.741, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 1.326, 95% CI 2-sided [-6.54 to 9.19]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300 mg; Test type: Superiority or Other; p = 0.983, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 0.083, 95% CI 2-sided [-7.76 to 7.93]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.041, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 8.204, 95% CI 2-sided [0.34 to 16.07]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10 mg; Test type: Superiority or Other; p = 0.475, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 2.891, 95% CI 2-sided [-5.05 to 10.83]

5. Secondary Outcome: Mean Change From Baseline in the Percentage of Symptom-free Nights Averaged Over the 8-Week Treatment Period
Description: Asthma symptoms were recorded in a daily eDairy by the participants every day in the morning upon rising and before taking any rescue or study medication and before the assessment of the PEF measurement. Participant's responses to the morning assessments indicated no symptoms were considered to be symptom free. For participants, the symptom free nights were assessed during the 8-Week treatment period. Change from Baseline was calculated as the averaged of symptom-free nights during the 8-Week treatment period minus the Baseline value (defined as the last 7 days prior to randomization of the participants).
Time Frame: Baseline up to Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free nights
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 30 mg | GSK2190915 100 mg | GSK2190915 300 mg | Fluticasone Propionate 100 mcg | Montelukast 10 mg
Number analyzed (Participants) | 99 | 99 | 99 | 100 | 101 | 100 | 97
Percentage of symptom-free nights | 13.99 (2.90) | 14.83 (2.90) | 16.71 (2.90) | 16.12 (2.88) | 12.21 (2.86) | 19.94 (2.88) | 19.39 (2.93)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; Test type: Superiority or Other; p = 0.838, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 0.837, 95% CI 2-sided [-7.22 to 8.89]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30 mg; Test type: Superiority or Other; p = 0.508, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 2.715, 95% CI 2-sided [-5.33 to 10.76]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100 mg; Test type: Superiority or Other; p = 0.603, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 2.124, 95% CI 2-sided [-5.90 to 10.14]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300 mg; Test type: Superiority or Other; p = 0.662, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Cox Proportional Hazard = -1.781, 95% CI 2-sided [-9.78 to 6.22]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.146, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 5.949, 95% CI 2-sided [-2.08 to 13.98]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10 mg; Test type: Superiority or Other; p = 0.191, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 5.394, 95% CI 2-sided [-2.69 to 13.48]

6. Secondary Outcome: Mean Change From Baseline in the Percentage of Rescue-free Days Averaged Over the 8-Week Treatment Period
Description: The number of inhalations of rescue salbutamol/albuterol inhalation aerosol used during the day and night was recorded by the participants in an eDiary. The time span during which the participants did not have to take any rescue medication (medication intended to relieve symptoms immediately) was considered to be a rescue-free period. For participants, the rescue-free days were assessed during the 8-Week treatment period. Change from Baseline was calculated as the averaged of rescue-free days during the 8-Week treatment period minus the Baseline value (defined as the last 7 days prior to randomization of the participants).
Time Frame: Baseline up to Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free days
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 30 mg | GSK2190915 100 mg | GSK2190915 300 mg | Fluticasone Propionate 100 mcg | Montelukast 10 mg
Number analyzed (Participants) | 99 | 99 | 99 | 100 | 101 | 101 | 97
Percentage of rescue-free days | 16.80 (3.10) | 22.91 (3.1) | 20.91 (3.09) | 18.95 (3.08) | 18.51 (3.06) | 26.39 (3.06) | 23.55 (3.13)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; Test type: Superiority or Other; p = 0.164, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 6.106, 95% CI 2-sided [-2.50 to 14.71]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30 mg; Test type: Superiority or Other; p = 0.349, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 4.106, 95% CI [-4.49 to 12.70]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100 mg; Test type: Superiority or Other; p = 0.623, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 2.148, 95% CI 2-sided [-6.42 to 10.72]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300 mg; Test type: Superiority or Other; p = 0.694, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 1.713, 95% CI 2-sided [-6.84 to 10.26]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.028, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 9.592, 95% CI 2-sided [1.03 to 18.15]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10 mg; Test type: Superiority or Other; p = 0.125, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 6.750, 95% CI 2-sided [-1.89 to 15.38]

7. Secondary Outcome: Mean Change From Baseline in the Percentage of Rescue-free Nights Averaged Over the 8-Week Treatment Period
Description: The number of inhalations of rescue salbutamol/albuterol inhalation aerosol used during the day and night was recorded by the participants in an eDiary. The time span during which the participants did not have to take any rescue medication (medication intended to relieve symptoms immediately) was considered to be a rescue-free period. For participants, the rescue-free nights were assessed during the 8-Week treatment period. Change from Baseline was calculated as the averaged of rescue-free nights during the 8-Week treatment period minus the Baseline value (defined as the last 7 days prior to randomization of the participants).
Time Frame: Baseline up to Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free nights
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 30 mg | GSK2190915 100 mg | GSK2190915 300 mg | Fluticasone Propionate 100 mcg | Montelukast 10 mg
Number analyzed (Participants) | 99 | 99 | 99 | 100 | 101 | 100 | 97
Percentage of rescue-free nights | 16.93 (3.04) | 19.28 (3.04) | 17.36 (3.03) | 19.63 (3.02) | 15.71 (3.00) | 24.42 (3.02) | 20.54 (3.07)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; Test type: Superiority or Other; p = 0.585, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 2.346, 95% CI 2-sided [-6.09 to 10.78]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30 mg; Test type: Superiority or Other; p = 0.920, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 0.431, 95% CI 2-sided [-8.00 to 8.86]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100 mg; Test type: Superiority or Other; p = 0.528, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 2.702, 95% CI 2-sided [-5.70 to 11.11]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300 mg; Test type: Superiority or Other; p = 0.776, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -1.218, 95% CI 2-sided [-9.60 to 7.17]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.081, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 7.490, 95% CI 2-sided [-0.92 to 15.90]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10 mg; Test type: Superiority or Other; p = 0.403, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 3.611, 95% CI 2-sided [-4.87 to 12.09]

8. Secondary Outcome: Mean Change From Baseline in Day-time Asthma Symptom Score Over the 8-Week Treatment Period
Description: Participants recorded their day-time asthma symptom score in an eDiary each PM at bedtime and before taking any rescue or study medication and before assessing the PEF measurement during the 8-Week treatment period. Day-time asthma symptom scores, as: 0=no asthma symptoms, 1=one episode of short-time asthma symptoms, 2=two or more episodes of short-time asthma symptoms, 3=asthma symptoms occurring during most part of daytime without interference with daily life activities, 4=asthma symptoms occurring during most part of daytime with interference with daily life activities, 5=severe asthma symptoms that disable working or perform normal daily activities. Change from Baseline was calculated as the averaged of day-time asthma symptom score during the 8-Week treatment period minus the Baseline value (defined as the last 7 days prior to randomization of the participants).
Time Frame: Baseline up to Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Day-time symptom scores on a scale
Groups:
- GSK2190915 10mg: Participants received one tablet of 10 mg GSK2190915 orally QD and one tablet of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
Arm/Group | Placebo | GSK2190915 10mg | GSK2190915 30mg | GSK2190915 100mg | GSK2190915 300mg | Fluticasone Propionate 100 mcg | Montelukast 10mg
Number analyzed (Participants) | 99 | 99 | 99 | 100 | 101 | 101 | 97
Day-time symptom scores on a scale | -0.34 (0.06) | -0.34 (0.06) | -0.50 (0.06) | -0.36 (0.06) | -0.34 (0.06) | -0.43 (0.06) | -0.41 (0.06)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10mg; Test type: Superiority or Other; p = 0.951, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.005, 95% CI 2-sided [-0.17 to 0.16]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30mg; Test type: Superiority or Other; p = 0.043, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.166, 95% CI 2-sided [-0.33 to -0.01]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100mg; Test type: Superiority or Other; p = 0.734, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.028, 95% CI 2-sided [-0.19 to 0.13]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300mg; Test type: Superiority or Other; p = 0.972, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.003, 95% CI 2-sided [-0.16 to 0.16]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.238, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.097, 95% CI 2-sided [-0.26 to 0.06]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10mg; Test type: Superiority or Other; p = 0.360, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.075, 95% CI 2-sided [-0.24 to 0.09]

9. Secondary Outcome: Mean Change From Baseline in Night-time Asthma Symptom Score Over the 8-Week Treatment Period
Description: Participants recorded their night-time asthma symptom score in an eDiary each AM upon rising and before taking any rescue or study medication and before assessing the PEF measurement during the 8-Week treatment period. Night-time asthma symptom scores, as: 0=no asthma symptoms, 1= one awakening or waking early due to asthma symptoms, 2= two or more awakenings due to asthma symptoms (including waking early), 3= asthma symptoms almost prevented the participant from sleeping, 4= severe asthma symptoms completely prevented from sleeping. Change from Baseline was calculated as the averaged of night-time asthma symptom score during the 8-Week treatment period minus the Baseline value (defined as the last 7 days prior to randomization of the participants).
Time Frame: Baseline up to Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Night-time symptom scores on a scale
Arm/Group | Placebo | GSK2190915 10mg | GSK2190915 30mg | GSK2190915 100mg | GSK2190915 300mg | Fluticasone Propionate 100 mcg | Montelukast 10mg
Number analyzed (Participants) | 99 | 99 | 99 | 100 | 101 | 100 | 97
Night-time symptom scores on a scale | -0.23 (0.05) | -0.21 (0.05) | -0.33 (0.05) | -0.26 (0.05) | -0.22 (0.05) | -0.29 (0.05) | -0.32 (0.05)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10mg; Test type: Superiority or Other; p = 0.692, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 0.028, 95% CI 2-sided [-0.11 to 0.17]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30mg vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.176, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.096, 95% CI 2-sided [-0.24 to 0.04]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100mg; Test type: Superiority or Other; p = 0.768, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.021, 95% CI 2-sided [-0.16 to 0.12]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300mg; Test type: Superiority or Other; p = 0.887, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = 0.010, 95% CI 2-sided [-0.13 to 0.15]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.471, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.051, 95% CI 2-sided [-0.19 to 0.09]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10mg; Test type: Superiority or Other; p = 0.248, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.083, 95% CI 2-sided [-0.22 to 0.06]

10. Secondary Outcome: Mean Change From Baseline in Day-time Rescue Short Acting beta2-agonist (SABA) Usage Over the 8-Week Treatment Period
Description: The number of inhalations of rescue SABA, salbutamol/albuterol inhalation aerosol used during the day and night was recorded by the participants in an eDiary. Participants who used salbutamol/albuterol inhalation aerosol at day-time were assessed during the 8-Week treatment period. Change from Baseline was calculated as the averaged number of day-time salbutamol/albuterol inhalation aerosol used during the 8-Week treatment period minus the Baseline value (defined as the last 7 days prior to randomization of the participants).
Time Frame: Baseline up to Week
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Day-time number of inhalations
Arm/Group | Placebo | GSK2190915 10mg | GSK2190915 30mg | GSK2190915 100mg | GSK2190915 300mg | Fluticasone Propionate 100 mcg | Montelukast 10mg
Number analyzed (Participants) | 99 | 99 | 99 | 100 | 101 | 101 | 97
Day-time number of inhalations | -0.42 (0.07) | -0.55 (0.07) | -0.68 (0.07) | -0.50 (0.07) | -0.47 (0.07) | -0.67 (0.07) | -0.63 (0.07)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10mg; Test type: Superiority or Other; p = 0.209, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.131, 95% CI 2-sided [-0.33 to 0.07]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30mg; Test type: Superiority or Other; p = 0.011, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.264, 95% CI 2-sided [-0.47 to -0.06]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100mg; Test type: Superiority or Other; p = 0.464, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.076, 95% CI 2-sided [-0.28 to 0.13]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300mg; Test type: Superiority or Other; p = 0.662, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.045, 95% CI 2-sided [-0.25 to 0.16]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.018, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.245, 95% CI 2-sided [-0.45 to -0.04]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10mg; Test type: Superiority or Other; p = 0.047, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.207, 95% CI 2-sided [-0.41 to -0.00]

11. Secondary Outcome: Mean Change From Baseline in Night-time Rescue SABA Usage Over the 8-Week Treatment Period
Description: The numbers of inhalations of rescue SABA, salbutamol/albuterol inhalation aerosol used during the day and night was recorded by the participants in an eDiary. Participants who used salbutamol/albuterol inhalation aerosol at night-time were assessed during the 8-Week treatment period. Change from Baseline was calculated as the averaged number of night-time salbutamol/albuterol inhalation aerosol used during the 8-Week treatment period minus the Baseline value (defined as the last 7 days prior to randomization of the participants).
Time Frame: Baseline up to Week 8
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Night-time number of inhalations
Groups:
- GSK2190915 10 0mg: Participants received one tablet of 100 mg GSK2190915 orally QD and one tablet of placebo orally plus one dose of FP matching placebo BID via DPI in morning and another dose of FP matching placebo via DPI plus one capsule of montelukast matching placebo orally QD in evening for the 8-Weeks.
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 30 mg | GSK2190915 10 0mg | GSK2190915 300 mg | Fluticasone Propionate 100 mcg | Montelukast 10 mg
Number analyzed (Participants) | 99 | 99 | 99 | 100 | 101 | 100 | 97
Night-time number of inhalations | -0.30 (0.07) | -0.40 (0.07) | -0.44 (0.07) | -0.42 (0.07) | -0.30 (0.07) | -0.47 (0.07) | -0.46 (0.07)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; Test type: Superiority or Other; p = 0.300, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.098, 95% CI 2-sided [-0.28 to 0.09]
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30 mg; Test type: Superiority or Other; p = 0.145, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.138, 95% CI 2-sided [-0.32 to 0.05]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 10 0mg; Test type: Superiority or Other; p = 0.190, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.123, 95% CI 2-sided [-0.31 to 0.06]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300 mg; Test type: Superiority or Other; p = 0.980, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.002, 95% CI 2-sided [-0.19 to 0.18]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.070, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.171, 95% CI 2-sided [-0.36 to 0.01]
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10 mg; Test type: Superiority or Other; p = 0.095, ANCOVA; Analysis was performed using ANCOVA with covariates of Baseline, age, gender, country and smoking status; Mean Difference (Net) = -0.158, 95% CI 2-sided [-0.34 to 0.03]

12. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy During the 8-Week Treatment Period
Description: The participants who met any of the following withdrawal criteria were considered to be withdrawn due to lack of efficacy: 1) Clinic FEV1 below stability limit calculated at Visit 3. 2) More than three days between two consecutive visits, PEF has fallen below stability limit calculated at Visit 3. 3) Use of 12 or more inhalations of SABA per day for more than two days between consecutive visits. 4) Asthma exacerbation defined as worsening requiring any treatment other than study medication or rescue medication. This included requiring the use of systemic or inhaled corticosteroids and /or emergency room visit or hospitalization for the treatment of asthma. The stability limit was calculated as best pre-salbutamol/albuterol FEV1 at Visit 3 x 80 percent (%).
Time Frame: Upto 8 Weeks
Population: ITT Population. Only those participants with analyzable data at the indicated time point were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2190915 10mg | GSK2190915 30mg | GSK2190915 100mg | GSK2190915 300mg | Fluticasone Propionate 100 mcg | Montelukast 10mg
Number analyzed (Participants) | 100 | 99 | 100 | 100 | 101 | 103 | 97
Participants | 11 | 11 | 9 | 11 | 13 | 8 | 7
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10mg; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 30mg; Test type: Superiority or Other; p = 0.814, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100mg; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 300mg; Test type: Superiority or Other; p = 0.828, Fisher Exact
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Propionate 100 mcg; Test type: Superiority or Other; p = 0.477, Fisher Exact
Statistical Analysis 6: Comparison: Placebo vs Montelukast 10mg; Test type: Superiority or Other; p = 0.460, Fisher Exact

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of administration of the study drug until the follow-up contact (up to Week 9).
Description: SAEs and non-serious AEs were reported for members of the ITT population.
Arm/Group | Placebo | GSK2190915 10mg | GSK2190915 30mg | GSK2190915 100mg | GSK2190915 300mg | Fluticasone Propionate 100 mcg | Montelukast 10mg
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/99 | 0/100 | 0/100 | 0/101 | 0/103 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/99 | 0/100 | 1/100 | 0/101 | 1/103 | 0/97
Other Adverse Events (participants affected / at risk) | 10/100 | 13/99 | 6/100 | 9/100 | 9/101 | 14/103 | 15/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | GSK2190915 10mg (N=99) | GSK2190915 30mg (N=100) | GSK2190915 100mg (N=100) | GSK2190915 300mg (N=101) | Fluticasone Propionate 100 mcg (N=103) | Montelukast 10mg (N=97)
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | GSK2190915 10mg (N=99) | GSK2190915 30mg (N=100) | GSK2190915 100mg (N=100) | GSK2190915 300mg (N=101) | Fluticasone Propionate 100 mcg (N=103) | Montelukast 10mg (N=97)
Headache (Nervous system disorders) | 3 | 7 | 2 | 4 | 4 | 9 | 9
Nasopharyngitis (Infections and infestations) | 5 | 6 | 3 | 2 | 5 | 5 | 5
Pharyngitis (Infections and infestations) | 2 | 0 | 1 | 3 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.